CLINICAL TRIAL: NCT04040595
Title: The Genetics of Adipose Tissue Function and Its Link to Type 2 Diabetes and Heart Disease
Acronym: FATFUNgenes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); NIHR Exeter Clinical Research Facility (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRAS: 257693; 105009 (Other Grant/Funding Number: Diabetes UK); 19/SW/0012 (Other: South West - Central Bristol Research Ethics Committee); 1909872 (Other: The Royal Devon & Exeter NHS Foundation Trust)
Record Dates: First submitted 2019-06-12; First posted 2019-07-31 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 diabetes; adipocyte; adipocyte tissue dysfunction; adiposity; favourable adiposity; gene expression; adipose tissue
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Anthropometry:
  * Baseline data including Height (m), Weight (kg), Waist (cm) and Hip (cm) circumference will be recorded.
  * Skin fold measurements (mm) from biceps, triceps, subscapular, and suprailiac regions
  * Detailed body fat measures will be obtained from the BodPodTM.
  Medical history:
  • including current medications and lifestyle information (smoking/alcohol).
  Blood sample:
  • Up to 20 ml venous blood sample for HbA1c and storage for analysis of biomarkers of adiposity.
  Abdominal fat biopsy: for adipocyte measurements and store a sample for future analyses.
  A sample of abdominal fat will be obtained by firstly injecting some local anaesthetic into an accessible area of the abdomen. Using a scalpel, a small incision (approx 2-3 cm) will be made to a depth of approx15mm and two small pea-sized samples of fat will be removed. The wound will be closed with simple sutures or steristrips.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adipocyte measurement (Experimental): Abdominal fat biopsy
  Interventions: Procedure: Abdominal fat biopsy

INTERVENTIONS:
Procedure: Abdominal fat biopsy — A sample of abdominal fat will be obtained by firstly injecting some local anaesthetic into an accessible area of the abdomen. Using a scalpel, a small incision (approx 2-3 cm) will be made to a depth of approx 15mm and two small pea-sized samples of fat will be removed. The wound will be closed with simple sutures or steristrips.

SUMMARY:
Obesity is a major risk factor for Type 2 diabetes. However, two obese people of the same height and weight can have very different risks of the condition. As a greater proportion of the population is becoming obese, scientists need to understand more about why some people develop Type 2 diabetes at lower weight and why some people stay healthy despite being obese. The investigators and others provided evidence for genetic factors associated with higher weight for a given height but lower risk of diabetes, lower cholesterol and fat levels, lower blood pressure and lower risk of heart disease. The investigators showed that people who carry these genetic factors are able to store extra fat in a safe place, which is under the skin, as they gain weight. The proposed project aims to establish whether or not these genetic factors are associated with better development and function of fat tissue in storing extra fat. It is thought that a healthy and functional fat tissue in the human body has a key role in modifying the risk of diseases such as Type 2 diabetes, heart disease and hypertension.

Volunteers from Exeter 10,000 who gave their permission to contact them about further research will be recruited to the study. In those that agree, detailed body size measures, including body composition assessments by the BodPodTM machine will be recorded, a blood sample will be collected, and a small subcutaneous abdominal fat biopsy will be collected to measure fat cell size and from which a sample will be stored for future analyses. The results between people with and without the particular genetic changes of interest will be compared.

Knowing more about these genetic changes and how fat cells work could help to improve understanding of the factors that predispose, delay or protect obese individuals from Type 2 diabetes and other metabolic disturbances.

DETAILED DESCRIPTION:
Introduction:

Diabetes is the most common chronic metabolic disease and is a major source of morbidity and mortality. It is one of the biggest healthcare challenges facing the United Kingdom's (UK) National Health Service (NHS) with more than 2.6 million adults diagnosed in the UK, with the vast majority (90%) having Type 2 diabetes (T2D). It is anticipated that the numbers will continue to rise, in part due to the increasing levels of obesity in the population.

Type 2 diabetes is characterised by high blood glucose levels in the context of increasing insulin resistance and reduced beta cell function, and this can develop over several years with individuals unaware of the problem.

Research groups in Exeter are leading efforts to identify the genetic factors that influence why some people develop Type 2 diabetes despite relative leanness, whilst many obese people do not get the disease. The investigators have identified many such factors but now wish to study them in more detail to understand the role of a healthy and functioning adipose tissue in the disease mechanism. This study builds on a previous 'recruit by genotype' study to explore the size of fat cells in people carrying the most genetic factors for being fatter but healthier (fATDIVA (for Adipose Tissue DIabetes VAriants) NCT02505321). The investigators will expand on the range of genetic variations to be undertaken in the research volunteers. The preliminary data from fATDIVA helped to secure prestigious funding from Diabetes UK to expand this work to improve understanding of the complex processes that lead to Type 2 diabetes.

The investigators are trying to understand how genetic variations cause differences in the human ability to store fat. The hypothesis to be tested is that individuals carrying different genetic variations have different abilities to store fat under the skin as subcutaneous fat tissue. This could lead to an improved understanding of subcutaneous fat storage. It is very unlikely that scientists will be able to reverse substantially the rising numbers of people becoming overweight or obese as they age, therefore this study's findings could be important in identifying how to reduce the risk of disease caused by obesity.

Study Design:

This is a prospective observational study that will take place over a 30 month period (March 2019 to August 2021).

Study participants:

All participants will be identified from existing research cohorts managed by the National Institute for Health Research (NIHR) Exeter Clinical Research Facility (Exeter CRF) and recruitment will be facilitated within the Exeter CRF.

Under over-arching ethical approval 09/H0106/75, approximately 8900 anonymised DNA samples have whole genome genotype data.

Subject Selection:

The researchers will provide the Exeter Clinical Research Facility (Exeter CRF) with a list of the sample numbers that fulfil the inclusion criteria. The Exeter CRF will approach these individuals on the researcher's behalf to ask if they would be willing to provide body fat measures, a blood sample and an abdominal fat biopsy. Participants would be invited to a single visit lasting up to 2 hours at the Exeter CRF for data and sample collection.

Interested participants will then be contacted directly by a member of the study team who will be responsible for the recruitment process, providing more detailed verbal and written project-specific information.

The investigators will aim to target men only to increase power for two reasons. First, men and women have different body shape and different fat distribution. Men tend to store the extra fat in abdominal subcutaneous adipose tissue while women tend to store it in the lower body. Second, the study of fat biopsy samples in women could be affected by menopause which could cause bias in the data.

However, as the target sample size is 500 and the number of men who fulfil the inclusion criteria is approximately 3000, this will be reviewed after a year. If projections indicate that the target sample size will not be met, women will also be recruited in the second year.

ELIGIBILITY:
Inclusion Criteria:

* Demographics: Age 18-75 inclusive
* Ethnicity: Reflective of local demographic
* Mental capacity: Willing and able to provide informed consent

Exclusion Criteria:

* Medical history: History of bariatric surgery and recent significant weight loss/gain (+/- 3 kgs/ half a stone in the last 3 months); connective tissue disease, pregnancy and lactation (if women are recruited).
* Medications: Currently prescribed oral/IV corticosteroid treatment or loop diuretics (furosemide, bumetanide), antiplatelet and anticoagulation medication, methotrexate
* Mental capacity: Unable/unwilling to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Mean adipocyte size (µm2) assessed using Image J software. | Within 12 months of recruitment date of final participant
  ImageJ is a cross-platform image analysis tool developed to measure particle/cell size and will be used here to measure adipocyte size to test whether or not individuals carrying a high genetic load of "favourable adiposity" alleles have smaller subcutaneous fat cells.

SECONDARY OUTCOMES:
Adipose tissue expression of genes that are markers of adipogenesis (PPARy, CREBP). | Within 12 months of recruitment date of final participant
  This secondary outcome is the adipocytes' gene expression measures of adipogenesis.
Adipose tissue expression of genes that are markers of fibrosis (SPARC, collagens, TGFbeta, LOX). | Within 12 months of recruitment date of final participant
  This secondary outcome is the adipocytes' gene expression measures of fibrosis.
Adipose tissue expression of genes that are determinants of adipose inflammation (IL-1beta, IL-6, and 8, TNFalpha, MCP-1/CCL2). | Within 12 months of recruitment date of final participant
  This secondary outcome is the adipocytes' gene expression measures of adipose inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Frayling, PhD, Principal Investigator — University of Exeter
Locations (1):
- Royal Devon and Exeter NHS Foundation Trust / University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruderman N, Chisholm D, Pi-Sunyer X, Schneider S. The metabolically obese, normal-weight individual revisited. Diabetes. 1998 May;47(5):699-713. doi: 10.2337/diabetes.47.5.699. PMID 9588440
- [Background] Ruderman NB, Schneider SH, Berchtold P. The "metabolically-obese," normal-weight individual. Am J Clin Nutr. 1981 Aug;34(8):1617-21. doi: 10.1093/ajcn/34.8.1617. PMID 7270486
- [Background] Ji Y, Yiorkas AM, Frau F, Mook-Kanamori D, Staiger H, Thomas EL, Atabaki-Pasdar N, Campbell A, Tyrrell J, Jones SE, Beaumont RN, Wood AR, Tuke MA, Ruth KS, Mahajan A, Murray A, Freathy RM, Weedon MN, Hattersley AT, Hayward C, Machann J, Haring HU, Franks P, de Mutsert R, Pearson E, Stefan N, Frayling TM, Allebrandt KV, Bell JD, Blakemore AI, Yaghootkar H. Genome-Wide and Abdominal MRI Data Provide Evidence That a Genetically Determined Favorable Adiposity Phenotype Is Characterized by Lower Ectopic Liver Fat and Lower Risk of Type 2 Diabetes, Heart Disease, and Hypertension. Diabetes. 2019 Jan;68(1):207-219. doi: 10.2337/db18-0708. Epub 2018 Oct 23. PMID 30352878
- [Background] Yaghootkar H, Lotta LA, Tyrrell J, Smit RA, Jones SE, Donnelly L, Beaumont R, Campbell A, Tuke MA, Hayward C, Ruth KS, Padmanabhan S, Jukema JW, Palmer CC, Hattersley A, Freathy RM, Langenberg C, Wareham NJ, Wood AR, Murray A, Weedon MN, Sattar N, Pearson E, Scott RA, Frayling TM. Genetic Evidence for a Link Between Favorable Adiposity and Lower Risk of Type 2 Diabetes, Hypertension, and Heart Disease. Diabetes. 2016 Aug;65(8):2448-60. doi: 10.2337/db15-1671. Epub 2016 Apr 26. PMID 27207519
- [Background] Yaghootkar H, Scott RA, White CC, Zhang W, Speliotes E, Munroe PB, Ehret GB, Bis JC, Fox CS, Walker M, Borecki IB, Knowles JW, Yerges-Armstrong L, Ohlsson C, Perry JR, Chambers JC, Kooner JS, Franceschini N, Langenberg C, Hivert MF, Dastani Z, Richards JB, Semple RK, Frayling TM. Genetic evidence for a normal-weight "metabolically obese" phenotype linking insulin resistance, hypertension, coronary artery disease, and type 2 diabetes. Diabetes. 2014 Dec;63(12):4369-77. doi: 10.2337/db14-0318. Epub 2014 Jul 21. PMID 25048195
- [Background] Lotta LA, Gulati P, Day FR, Payne F, Ongen H, van de Bunt M, Gaulton KJ, Eicher JD, Sharp SJ, Luan J, De Lucia Rolfe E, Stewart ID, Wheeler E, Willems SM, Adams C, Yaghootkar H; EPIC-InterAct Consortium; Cambridge FPLD1 Consortium; Forouhi NG, Khaw KT, Johnson AD, Semple RK, Frayling T, Perry JR, Dermitzakis E, McCarthy MI, Barroso I, Wareham NJ, Savage DB, Langenberg C, O'Rahilly S, Scott RA. Integrative genomic analysis implicates limited peripheral adipose storage capacity in the pathogenesis of human insulin resistance. Nat Genet. 2017 Jan;49(1):17-26. doi: 10.1038/ng.3714. Epub 2016 Nov 14. PMID 27841877
- [Background] Scott RA, Fall T, Pasko D, Barker A, Sharp SJ, Arriola L, Balkau B, Barricarte A, Barroso I, Boeing H, Clavel-Chapelon F, Crowe FL, Dekker JM, Fagherazzi G, Ferrannini E, Forouhi NG, Franks PW, Gavrila D, Giedraitis V, Grioni S, Groop LC, Kaaks R, Key TJ, Kuhn T, Lotta LA, Nilsson PM, Overvad K, Palli D, Panico S, Quiros JR, Rolandsson O, Roswall N, Sacerdote C, Sala N, Sanchez MJ, Schulze MB, Siddiq A, Slimani N, Sluijs I, Spijkerman AM, Tjonneland A, Tumino R, van der A DL, Yaghootkar H; RISC study group; EPIC-InterAct consortium; McCarthy MI, Semple RK, Riboli E, Walker M, Ingelsson E, Frayling TM, Savage DB, Langenberg C, Wareham NJ. Common genetic variants highlight the role of insulin resistance and body fat distribution in type 2 diabetes, independent of obesity. Diabetes. 2014 Dec;63(12):4378-4387. doi: 10.2337/db14-0319. Epub 2014 Jun 19. PMID 24947364
- [Background] Alkhouli N, Mansfield J, Green E, Bell J, Knight B, Liversedge N, Tham JC, Welbourn R, Shore AC, Kos K, Winlove CP. The mechanical properties of human adipose tissues and their relationships to the structure and composition of the extracellular matrix. Am J Physiol Endocrinol Metab. 2013 Dec;305(12):E1427-35. doi: 10.1152/ajpendo.00111.2013. Epub 2013 Oct 8. PMID 24105412
- [Background] Acosta JR, Douagi I, Andersson DP, Backdahl J, Ryden M, Arner P, Laurencikiene J. Increased fat cell size: a major phenotype of subcutaneous white adipose tissue in non-obese individuals with type 2 diabetes. Diabetologia. 2016 Mar;59(3):560-70. doi: 10.1007/s00125-015-3810-6. Epub 2015 Nov 25. PMID 26607638